CLINICAL TRIAL: NCT05951881
Title: Comparative Study Between a Pharmacy Technician and a Pharmacist in the Performance of Medication Anamneses in Emergency Departments: a Skills Validation Study
Brief Title: Comparative Study of the Performance of Drug Anamneses in an Emergency Department
Acronym: ProtocoleV4
Status: Completed | Type: Observational
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmacie - Protocole V4
Record Dates: First submitted 2023-03-20; First posted 2023-07-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urgent care unit patients with medication: All patients admitted to the emergency department who agree to describe their medication
  Interventions: Other: Emergency Care Unit - medicines

INTERVENTIONS:
Other: Emergency Care Unit - medicines — The same group of patients admitted to the emergency room will respond separately to a pharmacist and a pharmacy assistant about their daily medication.
  The two medical records will be compared in order to evaluate the work of the pharmacy assistant on the basis of 3 sources :
  * the Electronic Medical Record
  * the patient's medication history
  * the reference pharmacy

SUMMARY:
After the first medical history by the nurse and the emergency physician, the pharmacist and the pharmacy assistant take a detailed history of the patient's medications separately.

After checking with the patient's reference pharmacy, the pharmacist and pharmacy assistant compare their results.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the emergency care unit
* Over 18 years old
* Giving consent to participate

Exclusion Criteria:

* Patients who do not take medication daily
* Unconscious patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research is aimed at patients admitted to the emergency department of the Saint-Joseph site.
  All patients over 18 years of age who are capable of giving informed consent and who are taking several medications prior to their admission to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of identical medication anamneses between pharmacist and pharmacy assistant | immediately after admission to the emergency department
  A pharmacist and a pharmacy assistant will compare the medication history of all patients who meet the eligibility criteria

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Rosart, Pharmacist, Principal Investigator — Grand Hôpital de Charleroi
Locations (1):
- GHdC, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No